CLINICAL TRIAL: NCT04738292
Title: A Phase II Trial of OnapriStone in CoMbInation With FuLvestrant for Patients With ER-positive, and HER2-negative Metastatic Breast Cancer After Progression on Endocrine Therapy and CDK 4/6 Inhibitors
Brief Title: Onapristone and Fulvestrant for ER+ HER2- Metastatic Breast Cancer After Endocrine Therapy and CDK4/6 Inhibitors (The SMILE Study)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: funding
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Context Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UW20037; A534260 (Other: UW Madison); SMPH/MEDICINE/HEM-ONC (Other: UW Madison); 2020-0877 (Other: Institutional Review Board); NCI-2021-00371 (Registry Identifier: NCI CTRP); Protocol Version 8/26/2021 (Other: UW Madison)
Record Dates: First submitted 2021-02-01; First posted 2021-02-04 (Actual); Results first posted 2024-05-03 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-05

CONDITIONS: ER-positive Breast Cancer; HER2-negative Breast Cancer; Metastatic Cancer
MeSH Terms: conditions — Neoplasm Metastasis | interventions — onapristone; Fulvestrant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Onapristone In Combination with Fulvestrant (Experimental): All participants will receive onapristone 50 mg p.o. BID (twice) daily and fulvestrant (500 mg) intramuscular injection on days 1, 15 (cycle 1), then two weeks later (cycle 2, day1), then once every 28 days thereafter. A cycle is defined as 28 days.
  There will be no breaks between dosing cycles.
  Interventions: Drug: Onapristone; Drug: Fulvestrant

INTERVENTIONS:
Drug: Onapristone — Onapristone is a type I antiprogestin which prevents the PgR from dimerizing and blocks ligand induced protein kinase-mediated phosphorylation of the PgR.
Drug: Fulvestrant — Fulvestrant binds, blocks and degrades the ER, completely inhibiting ER signaling.
  Other Names: Fulvestrant Injection

SUMMARY:
A phase II single-arm trial of onapristone in combination with fulvestrant for women and men with ER-positive, PgR-positive or negative and HER2-negative locally advanced or metastatic breast cancer after progression on aromatase and CDK4/6 inhibitors. The study will enroll up to 39 participants.

ELIGIBILITY:
Inclusion Criteria:

* Advanced ER+, (PgR positive or negative), and HER2 negative breast cancer. Advanced is defined as locally advanced or locoregionally recurrent or metastatic and not amenable to curative therapy.
* Below-mentioned prior lines of therapy are allowed in the adjuvant and or metastatic ER+/HER2- setting.

  * Participants must have had prior endocrine therapy either in the adjuvant or metastatic setting (SERM (tamoxifen, raloxifene, toremifene) or any of the aromatase inhibitors (anastrozole, letrozole, exemestane), or oral selective estrogen receptor degrader (SERD) on a clinical trial either in the adjuvant or metastatic setting
  * Participants must have received prior therapy with oral cyclin-dependent kinase (CDK)4/6 inhibitors in the metastatic setting
  * Other standard therapies in the metastatic setting (such as mTOR inhibitors) are allowed
  * Patients who previously received any one of the standard adjuvant chemotherapy regimens in a curative setting are eligible for this study.
  * One line of prior chemotherapy in the metastatic setting is allowed (i.e. any single agent or doublet cytotoxic chemotherapy, not limited to xeloda).
* Histologically and/or cytologically confirmed diagnosis of ER+, PgR+/- and HER2- breast cancer by local laboratory at diagnosis of metastatic disease. Hormone receptor positivity is defined as ER and PgR positivity in at least 1% cells by immunohistochemistry (IHC). HER2-negative breast cancer is defined as a negative in situ hybridization test or an IHC status of 0, 1+ or 2+. If IHC is 2+, a negative in situ hybridization test is required.
* Measurable disease, i.e., at least one measurable lesion, as per RECIST 1.1 criteria. A palpable, and measurable breast mass is acceptable.
* Eastern Cooperative Oncology Group (ECOG) Performance status ≤ 2
* Adequate organ function as defined by

  * aspartate aminotransferase (AST), alanine aminotransferase (ALT) ≤ 2.5 times institutional upper limit.
  * Total bilirubin ≤ 1.5 × upper limit of normal (ULN), except for subjects with Gilbert's syndrome who may be included if their total bilirubin is ≤ 3.0 × ULN and direct bilirubin ≤ 1.5 × ULN.
  * Alkaline phosphatase (ALP) ≤ 2.5 times institutional upper limit with exception that ALP of < 5 x ULN is acceptable in patients with elevated with ALP due to bone metastases (in the absence of liver metastases).
  * Serum creatinine <1.5 × ULN.
  * Absolute neutrophil count (ANC) ≥1000/µL.
  * Participants with lymphopenia are eligible at the discretion of the treating provider
  * Hemoglobin (Hb) ≥ 8g/dL.
  * Platelet count ≥ 100,000/µL
* Female participants must meet one of the following:

  * Postmenopausal for at least one year before enrollment, or
  * Surgically sterile (i.e., undergone bilateral oophorectomy), or
  * Premenopausal is defined as someone who has had menses at any time in the preceding 12 months. Premenopausal women who are eligible for this trial will require a Gonadotropin-releasing hormone (GnRH) analogue and treating physician may choose to monitor the ovarian function with laboratory tests to ensure a complete menopausal status with cessation of menses
* Women of childbearing potential must have a negative pregnancy test within seven days of registration. Participants must have a negative pregnancy test seven to 10 days prior to starting study treatment
* A formalin fixed paraffin embedded (FFPE) tumor biopsy block or up to 20 superplus frost slides with unstained histological sections at 4 micrometer thickness are required at the time of study entry. Archived tumor tissue acceptable (metastatic disease from non-bone and non-brain sites preferred, but primary breast or lymph node tissue is permitted) if obtained in the 18 months prior to study registration, otherwise a fresh biopsy will be required if deemed safe by the treating physician (minimal risk to patient). Confirmation of adequate and available tissue sample is to be determined by the site's pathologist. Tumor samples do not need to be shipped for eligibility purposes. Tumor samples do not need to be shipped until subject is confirmed eligible and is registered for treatment.
* Ability to take oral medications (without crushing). Please refer to section 6.1.2 for directions on taking the study drug (onapristone).
* To participate in the optional 18F-FFNP PET/CT imaging, the subject must have ER positive, HER2 negative, AND PgR positive disease and at least one extra hepatic lesion measuring at least 10 mm in size.

Exclusion Criteria:

* Prior treatment with an anti-progesterone agent.
* Prior treatment with fulvestrant in the metastatic setting
* Prior treatment with CDK4/6 inhibitors in the neoadjuvant/adjuvant setting
* History of malignancy other than breast cancer within three years prior to registration except for adequately treated non-melanoma skin cancer, cervical carcinoma in situ.
* History or presence of clinically active, and symptomatic central nervous system (CNS) metastasis: If the patient fulfills the following criteria, they will be eligible for the trial:

  * Completed prior therapy (including radiation and/or surgery) for CNS metastases ≥ 28 days prior to the start of study treatment and CNS tumor is clinically stable at the time of screening and patient is not receiving steroids and/or enzyme inducing anti-epileptic medications for brain metastases.
* Participants with any of the following conditions:

  * Clinically significant illness or systemic disease as determined by the treating physicians.
  * Active hepatitis or uncontrolled infection or any other clinically significant cirrhosis or other disease that, in the opinion of the investigator would pose a risk to subject safety or interfere with the study evaluation, procedures or completion. Testing for infectious hepatitis is not required for the study. Treating provider may choose additional testing if indicated clinically.
* Patients who have had systemic chemotherapy, or targeted therapy, within two weeks prior to starting study treatment or those who have not recovered from acute effects of any prior therapy to baseline or Grade ≤1. Grade 2 or higher exceptions include alopecia, up to grade 2 neuropathy or other grade 2 adverse events (AEs) or lab values not constituting a safety risk in the pinion of the treating physician. NCI CTCAE v5.0 will be used.
* Co-administration with any prescriptions during the four weeks prior to first onapristone dosing and concerns for possible drug interactions should be discussed with the pharmacist
* Patients who are pregnant or breast feeding
* History of acute coronary syndromes (including myocardial infarction, unstable angina, coronary artery bypass grafting, coronary angioplasty, or stenting) or symptomatic pericarditis within 6 months prior to registration..
* Symptomatic congestive heart failure (New York Heart Association III-IV)
* Clinically significant cardiac arrhythmias (e.g. ventricular tachycardia), complete left bundle branch block, high-grade atrioventricular block (AV) block (e.g. bifascicular block, Mobitz type II and third-degree AV block).
* Any episode of atrial fibrillation in the prior 12 months.
* QT interval >480 msec.
* Long QT syndrome or family history of idiopathic sudden death or congenital long QT syndrome.
* Concomitant use of medication(s) with a known risk to prolong the QT interval and/or known to cause Torsades de Pointe that cannot be discontinued (within 5 half-lives or 7 days prior to starting study drug) or replaced by safe alternative medication.
* Systolic blood pressure (SBP) >160 mmHg or <90 mmHg at screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2021-10-05 (Actual); Primary Completion 2023-04-03 (Actual); Study Completion 2023-05-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kari B Wisinski, MD, Principal Investigator — University of Wisconsin, Madison; Sailaja Kamaraju, MD, MS, Study Chair — Medical College of Wisconsin
Locations (2):
- United States (2):
  - University of Wisconsin Carbone Cancer Center, Madison, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the UW Hospital and Clinics and the Medical College of Wisconsin between October 2021 and January 2023.
Groups:
- Onapristone In Combination With Fulvestrant: All participants will receive onapristone 50 mg p.o. BID (twice) daily and fulvestrant (500 mg) intramuscular injection on days 1, 15 (cycle 1), then two weeks later (cycle 2, day1), then once every 28 days thereafter. A cycle is defined as 28 days.
  There will be no breaks between dosing cycles.
  Onapristone: Onapristone is a type I antiprogestin which prevents the PgR from dimerizing and blocks ligand induced protein kinase-mediated phosphorylation of the PgR.
  Fulvestrant: Fulvestrant binds, blocks and degrades the ER, completely inhibiting ER signaling.
Period: Overall Study
Arm/Group | Onapristone In Combination With Fulvestrant
Started | 11
Completed | 10
Not Completed | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Arm/Group | Onapristone In Combination With Fulvestrant
Number analyzed (Participants) | 11
Age, Customized [Count of Participants; unit: Participants]
  30 to 39 years old | 1
  40 to 49 years old | 1
  50 to 59 years old | 3
  60 to 69 years old | 5
  70 to 79 years old | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 11
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Objective Response (ORR)
Description: Best overall response of complete response (CR) or partial response (PR), as per RECIST 1.1. Point and 95% interval estimate of ORR will be evaluated accounting for possibility of early futility stopping.
Time Frame: up to 17 months
Measure: Count of Participants; unit: Participants
Arm/Group | Onapristone In Combination With Fulvestrant
Number analyzed (Participants) | 11
Participants | 0

2. Secondary Outcome: Number of Participants Experiencing Progression Free Survival (PFS)
Description: Time from date of enrollment to the date of first documented disease progression or death due to any cause. PFS will be described with Kaplan-Meier (KM) Curve and its pointwise asymptotic 95% confidence bounds. Median PFS if reached will be extracted from this KM estimator.
Time Frame: up to 17 months
Measure: Count of Participants; unit: Participants
Arm/Group | Onapristone In Combination With Fulvestrant
Number analyzed (Participants) | 11
Participants
  1 year PFS | 0
  17 month PFS | 0

3. Secondary Outcome: Number of Participants With Disease Control (DCR)
Description: Best overall response of CR, PR or stable disease (SD) lasting for ≥ 24 weeks, as per RECIST 1.1. DCR will be estimated with relative frequency and exact two-sided 95% binomial confidence interval.
Time Frame: up to 17 months
Measure: Count of Participants; unit: Participants
Arm/Group | Onapristone In Combination With Fulvestrant
Number analyzed (Participants) | 11
Participants | 2

4. Secondary Outcome: Time to Response
Description: Time from registration to first documented response (CR or PR) will be evaluated with a cumulative incidence where death will be as a competing risk to response.
Time Frame: up to 17 months
Population: Time to response could not be calculated as there was not a response to treatment within the study time points.
Arm/Group | Onapristone In Combination With Fulvestrant
Number analyzed (Participants) | 0

5. Secondary Outcome: Duration of Response
Description: Time between the first date of documented response to progression or death due to breast cancer. Duration of response will be assessed for a subgroup of subjects with observed response. The date of response will be denoted as time zero and time to progression or death will be evaluated with KM curve and 95% confidence interval (CI). Median time to response will be extracted from this KM curve.
Time Frame: up to 17 months
Population: Duration of Response could not be calculated because there was no response to treatment within the study time points.
Arm/Group | Onapristone In Combination With Fulvestrant
Number analyzed (Participants) | 0

6. Secondary Outcome: Incidence of Treatment-Related Adverse Events
Description: Type, frequency and severity of adverse events and laboratory abnormalities (according to CTCAE version 5.0) will be summarized with descriptive frequency tables. See Adverse Events Section for detailed summary.
Time Frame: up to 17 months
Measure: Count of Participants; unit: Participants
Arm/Group | Onapristone In Combination With Fulvestrant
Number analyzed (Participants) | 11
Participants
  Participants Experiencing Grade 1 Adverse Events | 6
  Participants Experiencing Grade 2 Adverse Events | 1
  Participants Experiencing Grade 3 Adverse Events | 1

ADVERSE EVENTS:
Time Frame: from consent to 30 days following last dose of study drug (up to approximately 17 months)
Description: AEs may be spontaneously reported by the patient and/or in response to an open question from study personnel or revealed by observation, physical examination or other diagnostic procedures
Arm/Group | Onapristone In Combination With Fulvestrant
All-Cause Mortality (participants affected / at risk) | 1/11
Serious Adverse Events (participants affected / at risk) | 3/11
Other Adverse Events (participants affected / at risk) | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Onapristone In Combination With Fulvestrant (N=11)
Pain (General disorders) | 1 (1)
Lung Infection (Infections and infestations) | 1 (1)
Hip Fracture (Injury, poisoning and procedural complications) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Onapristone In Combination With Fulvestrant (N=11)
Fatigue (General disorders) | 4 (5)
Non-cardiac chest pain (General disorders) | 3 (3)
General disorders and administration site conditions - Other, specify (General disorders) | 1 (1) — Groin Pain
Chills (General disorders) | 1 (1)
Facial pain (General disorders) | 1 (1)
Fever (General disorders) | 1 (2)
Injection site reaction (General disorders) | 2 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 4 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (6)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 5 (5)
Nausea (Gastrointestinal disorders) | 4 (5)
Dry mouth (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 (1) — Loss of Appetite
Vomiting (Gastrointestinal disorders) | 2 (2)
Dizziness (Nervous system disorders) | 2 (2)
Headache (Nervous system disorders) | 3 (4)
Tremor (Nervous system disorders) | 1 (1)
Infections and infestations - Other, specify (Infections and infestations) | 1 (1) — COVID-19
Urinary tract infection (Infections and infestations) | 2 (2)
Fracture (Injury, poisoning and procedural complications) | 1 (3)
Anxiety (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 2 (2)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Blurred vision (Eye disorders) | 1 (1)
Flashing lights (Eye disorders) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 1 (1)
Urinary urgency (Renal and urinary disorders) | 1 (1)
Breast pain (Reproductive system and breast disorders) | 2 (2)
Gait Disturbance (General disorders) | 1 (1)
General disorders and administration site conditions - Other, specify (General disorders) | 1 (1) — Tooth Numbness
Flu like symptoms (General disorders) | 1 (1)
Muscle cramp (Musculoskeletal and connective tissue disorders) | 2 (2)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1 (1) — Muscle tightness
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Lymph node pain (Blood and lymphatic system disorders) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 1 (1) — Increased Blood Urea Nitrogen
Abdominal pain (Gastrointestinal disorders) | 4 (4)
Belching (Gastrointestinal disorders) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1)
Paresthesia (Nervous system disorders) | 1 (1)
Hypersomnia (Nervous system disorders) | 1 (1)
Memory impairment (Nervous system disorders) | 1 (1)
Delirium (Psychiatric disorders) | 1 (2)
Urinary incontinence (Renal and urinary disorders) | 2 (2)
Pelvic pain (Reproductive system and breast disorders) | 1 (1)
Hot flashes (Vascular disorders) | 2 (2)
Hypertension (Vascular disorders) | 4 (8)
Lymphedema (Vascular disorders) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 2 (2)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (2)
Hypoalbuminemia (Metabolism and nutrition disorders) | 3 (3)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Alanine aminotransferase increased (Investigations) | 3 (7)
Alkaline phosphatase increased (Investigations) | 3 (3)
Aspartate aminotransferase increased (Investigations) | 5 (7)
Blood bilirubin increased (Investigations) | 1 (1)
Lymphocyte count decreased (Investigations) | 3 (4)
Neutrophil count decreased (Investigations) | 1 (1)
Platelet count decreased (Investigations) | 1 (1)
White blood cell decreased (Investigations) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1)
Avascular necrosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Study was terminated early, sponsor closed study. Study not powered per protocol.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-26): https://cdn.clinicaltrials.gov/large-docs/92/NCT04738292/Prot_SAP_000.pdf